CLINICAL TRIAL: NCT00802659
Title: A Phase I/II Dose Escalation Study to Evaluate Pain Response Using Extracranial Stereotactic Radiosurgery to Treat Paraspinal Metastasis in Patients Who Have Received Prior Spinal Irradiation
Brief Title: A Phase I/II Dose Escalation Study Using Extracranial Stereotactic Radiosurgery to Control Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-1149
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group -1 (Experimental): 1000 cGY radiation
  Interventions: Radiation: Stereotactic radiotherapy
- Group 1 (Experimental): 1200 cGY radiation
  Interventions: Radiation: Stereotactic radiotherapy
- Group 2 (Experimental): 1400 cGY radiation
  Interventions: Radiation: Stereotactic radiotherapy
- Group 3 (Experimental): 1600 cGY radiation
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — This study has 4 treatment groups: This will be determined based on what radiation treatment doses have been previously given to the patient on this study, how effective the dose has been with treatment patient's pain, and how many side effects participants before you have experienced.
  Other Names: Stereotactic Radiosurgery; Paraspinal Metastasis; Prior Spinal Irradiation

SUMMARY:
This study will evaluate pain control and quality of life in patients with paraspinal metastases, who have receive previous radiation therapy to these lesions, using single dose stereotactic radiotherapy.

DETAILED DESCRIPTION:
The goal of the study is to determine the lowest dose of radiation that can be given to effectively control the tumor and provide effective pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Prior non-hematogenous, histologically proven malignancy (specific exclusions are multiple myeloma and lymphoma)
* Pain attributable to one or two radiographically apparent metastatic lesion(s) amenable to ESRT
* Have had prior radiation to area of spine felt to be cause of patient's pain
* Zubrod performance status of 0-3
* Life expectancy of ≥ 3 months
* Signed informed consent prior to registration to study
* Radiographic evidence of stable disease outside of the spinal column for at least 6 weeks prior to study entry, as evaluated by pre-study imaging.

Exclusion Criteria:

* Women who are pregnant or nursing
* Either 'no evidence of other active cancerous disease' or 'other sites of known disease are locally controlled'
* No radiographic evidence of spinal instability (e.g. spinal cord compression requiring immediate surgical intervention)
* No initiation of chemotherapy within 15 days of trial entry.
* No plans for concomitant antineoplastic therapy (including standard fractionated RT, chemotherapy, biologic, vaccine therapy, or surgery) for at least 15 days following stereotactic radiosurgery.
* No active systemic infection.
* No evidence of myelopathy or cauda equina syndrome on clinical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- See also: (AlvinJ. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Group -1: 1000 cGY radiation
  Stereotactic radiotherapy: This study has 4 treatment groups: This will be determined based on what radiation treatment doses have been previously given to the patient on this study, how effective the dose has been with treatment of patient's pain, and how many side effects participants before have experienced.
- Group 1: 1200 cGY radiation
  Stereotactic radiotherapy: This study has 4 treatment groups: This will be determined based on what radiation treatment doses have been previously given to the patient on this study, how effective the dose has been with treatment of patient's pain, and how many side effects participants before have experienced.
- Group 2: 1400 cGY radiation
  Stereotactic radiotherapy: This study has 4 treatment groups: This will be determined based on what radiation treatment doses have been previously given to the patient on this study, how effective the dose has been with treatment of patient's pain, and how many side effects participants before have experienced.
- Group 3: 1600 cGY radiation
  Stereotactic radiotherapy: This study has 4 treatment groups: This will be determined based on what radiation treatment doses have been previously given to the patient on this study, how effective the dose has been with treatment of patient's pain, and how many side effects participants before have experienced.
Period: Overall Study
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Started | 0 | 2 | 0 | 0
Completed | 0 | 1 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 |  |  | 0
  Between 18 and 65 years |  | 1 |  |  | 1
  >=65 years |  | 0 |  |  | 0
Gender [Number; unit: participants]
  Female |  | 1 |  |  | 1
  Male |  | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose of Stereotactic Spinal Irradiation Needed to Obtain Durable Pain Control at 4 Weeks in a Previously Irradiated Spine Field
Description: Optimal dose
  1. the maximum tolerated dose (MTD) that will result in a 10% ESRT-induced neurological complications
  2. the minimal dose level that can achieve an 80% or more pain control rate, whichever occurs first
Time Frame: 4 weeks
Population: Group 1 was the only group to have a participant enrolled; however this outcome was not measured because there was not enough participants enrolled to provide the needed data for analysis.
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Duration of Pain Control for Each Dose Level.
Description: A reduction in pain, referable to the site of the spine lesion, by >=30% according to the Brief Pain Inventory (BPI), or a smaller decrease in pain accompanied by a reduction of pain medications.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Determine the Rate of Radiation-induced Myelopathy From Stereotactic Re-irradiation of the Spinal Metastases.
Time Frame: 4 weeks
Population: as for outcome 1
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Determine the Pattern of Failure After Stereotactic Irradiation of Spinal Metastases.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Quality of Life
Description: As measured by the Functional Assessment of Cancer Therapy - Central Nervous System (FACT-CNS)
  Participant can chose on a scale of 0-4 with 0=not at all and 4=very much.
Time Frame: 4 years
Population: as for outcome 1
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group -1 | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group -1 (N=0) | Group 1 (N=1) | Group 2 (N=0) | Group 3 (N=0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Death NOS (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group -1 (N=0) | Group 1 (N=1) | Group 2 (N=0) | Group 3 (N=0)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Investigations) | 0 | 1 | 0 | 0
Platelets (Investigations) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was closed early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes